CLINICAL TRIAL: NCT04869215
Title: Effect of EverVita Pro, a Protein Rich Ingredient, on Satiety Measures, Subsequent Energy Intake, and Gastrointestinal Symptoms: A Randomized, Controlled, Cross-over Study in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evergrain, LLC (Industry)
Collaborators: INQUIS Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Satiety EVP in bread
Record Dates: First submitted 2021-04-29; First posted 2021-05-03 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Satiety of High Fiber High Protein Bread
Keywords: satiation, fullness, protein, fiber, hunger, bread

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EverVita Pro consumed at breakfast followed by an ad lib meal (Experimental): Before breakfast, a Motivation to Eat and a GI symptom questionnaire will be completed. They will then be given a standard breakfast which will include EverVita Pro bread, followed by an ad lib pizza meal 1.5h later. Subjects will be asked to fill out the VAS Motivation to Eat Questionnaire before being given the meal and at 10-minute intervals after they start consuming the test meal until they are given the ad lib pizza meal and 30 min after the start of the ad lib pizza meal.
  Interventions: Other: EverVita Pro
- Control consumed at breakfast followed by an ad lib meal. (Placebo Comparator): Before breakfast, a Motivation to Eat and a GI symptom questionnaire will be completed. They will then be given a standard breakfast which will include the control bread, followed by an ad lib pizza meal 1.5h later. Subjects will be asked to fill out the VAS Motivation to Eat Questionnaire before being given the meal and at 10-minute intervals after they start consuming the test meal until they are given the ad lib pizza meal and 30 min after the start of the ad lib pizza meal.
  Interventions: Other: Control bread

INTERVENTIONS:
Other: EverVita Pro — EverVita Pro is composed of barley and corn, grown and mechanically processed in Europe, with non-GMO grains.
  Arms: EverVita Pro consumed at breakfast followed by an ad lib meal
Other: Control bread — Bread baked with normal Bakers flour
  Arms: Control consumed at breakfast followed by an ad lib meal.

SUMMARY:
This study will explore the satiating effect of EverVita Pro when consumed at breakfast on subsequent food intake. On 2 separate days, subjects will consume in random order a test breakfast (bread, butter, jam), either containing containing EverVita Pro or not (control), followed by an ad libitum pizza lunch 1.5 hours later. Before breakfast, after breakfast and after the pizza, subjects will fill in questionnaires regarding their motivation to eat (feelings of hunger/fullness). The hypothesis is that the EverVita Pro breakfast will result in less pizza consumption and prolonged feeling of fullness and satiety in comparison to the control bread.

DETAILED DESCRIPTION:
A standard breakfast meal will be consumed at each visit and it will contain either the test (EverVita Pro) or control product. The test meals and control meals are designed to be isocaloric. The portion size of the EverVitaPro or Control bread is matched in the calories equivalent to 3 slices of wholemeal bread.

A (GI) symptoms questionnaire will be administered to assess GI tolerability: 1) before breakfast (0'), 2) before ad -libitum pizza lunch (90'), 3) before bedtime, and 4) before breakfast the following morning (24h). Comparison of satiety scores at each time point for each individual question between test and control over 2h. Subjective measurements of motivation to eat will be assessed using visual analog scales (VAS) by filling out the VAS motivation to eat questionnaire. For instance, fullness is assessed with the following statement on the left side of the line "not full at all" with the following statement to the right side of the line "As full as I have ever felt". Participants will place a vertical line along the horizontal line to the point that they feel reflects their feelings at that moment. Subjects will not be permitted to refer to their previous ratings when completing the VAS.

Power calculation was done for a two-sided, two-sample t-test assuming equal variances and equal sample sizes for the two groups to detect a 700 KJ difference in intake between products using a non-central t-distribution.

A sample size of 60 subjects, 30 per sequence, is sufficient to detect a 700 KJ difference in intake between products with 94% statistical power if the standard deviation for intake is as large as 1500 KJ.

Randomization Individuals are allocated to the two sequence of preloads (EverVita Pro meal/Control meal and Control meal/EverVita Pro meal) completely at random.

Statistical Analysis

Primary Objective:

The primary outcome (response) measured is the energy intake 90 min after preload administration.

Secondary Objectives:

Visual analogue scores (VAS) from 4 questions (Desire to eat, Hunger, Fullness, Prospective consumption) and gastrointestinal severity symptoms from 9 questions (Diarrhea, Vomiting, Abdominal distension, Hiccups, Stomach aches/abdominal pain, Constipation, Flatulence or gas in abdomen, Nausea, Indigestion) are evaluated as secondary outcomes.

Data are presented as mean ± SEM unless stated otherwise. All statistical analyses are performed using R statistical software, version 3.6.3 (http://www.r-project.org/). All test are two-sided and a value of P < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 30kg/m2, inclusive
* No major illness or surgery requiring hospitalization within 3 months of the screening visit
* Subjects must be eligible to receive income in Canada.
* Understanding Subjects must understand the study procedures and be willing to provide informed consent to participate in the study
* Individuals who are able to become pregnant are willing to avoid pregnancy during the study period

Exclusion Criteria:

* Failure to meet all the inclusion criteria
* Smokers (cigarettes, vape, cannabis)
* Pregnant or breastfeeding (self-reported)
* Known history of diabetes, liver disease, renal failure, gallstone disease, significant cardiovascular disease, major psychiatric disorders or other medical conditions which might, in the opinion of the Principal Investigator (PI), either 1) make participation dangerous to the subject or to others, 2) affect the results, or 3) influence the ability of the subject to comply with study procedures
* Use of any drug which would interfere with appetite, in the opinion of the PI.
* Unwillingness or inability to comply with the experimental procedures and to follow INQUIS safety guidelines
* Known intolerance, sensitivity or allergy to any ingredients in the study products
* History of cancer in the prior two years, except for non-melanoma skin cancer

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Energy intake comparison | at time point 1.5 hours
  Compare energy intake from the ad libitum pizza meal following the EverVita Pro containing meal and a control meal.

SECONDARY OUTCOMES:
Satiety scores from VAS per individual | every 10 minutes for 90 minutes, then after 120 minutes again
  Compare satiety scores at each time point for each individual question between EverVita Protest and control over 2h
Satiety scores from VAS between individuals | every 10 minutes for 90 minutes, then after 120 minutes again
  Compare composite satiety score at each time point between EverVita Pro and control over 2h
Gastrointestinal effects via GI symptoms questionnaire | at t=0, after 90 minutes, before bed time and 24 hours after start intervention
  Compare the incidence and severity of GI symptoms after ingestion of EverVita Pro with a control over 24h

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, DM, PhD, Principal Investigator — INQUIS Clinical Research
Locations (1):
- INQUIS Clinical Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No